CLINICAL TRIAL: NCT03778892
Title: Youth-focused Strategies to Promote Adherence to Pre-exposure Prophylaxis Among Youth At-risk for HIV in Thailand
Acronym: YouthPrEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Collaborators: Thai Red Cross AIDS Research Centre (Other); International AIDS Society (Other)
Responsible Party: Principal Investigator, Wipaporn Natalie Songtaweesin, MD., Principal Investigator, Clinical Researcher, Chulalongkorn University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2017/472-SON
Record Dates: First submitted 2018-12-08; First posted 2018-12-19 (Actual); Last update posted 2020-01-23 (Actual); Status verified 2020-01

CONDITIONS: Adherence, Medication; Adolescent Behavior; HIV Prevention; Sexual Health; Mobile Health
Keywords: PrEP adherence; Youth; Adolescents; MSM; HIV Prevention; Mobile Health
MeSH Terms: conditions — Medication Adherence; Adolescent Behavior

STUDY DESIGN:
Intervention Model Description: half of study participants will receive the intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Novel Intervention (Experimental): Use of a mobile phone application to support PrEP adherence in addition to youth-friendly counselling and services
  Interventions: Behavioral: 'Project Raincoat' Mobile Phone Application
- Standard Intervention (No Intervention): Use of a mobile phone application to support PrEP adherence in addition to youth-friendly counselling and services

INTERVENTIONS:
Behavioral: 'Project Raincoat' Mobile Phone Application — Mobile phone application with weekly input channels for PrEP use, condom use, number of sex partners and sex acts and a calculation of self-HIV risk feedback scoring. Scoring system for attendance of visits, normal blood tests and use of application. Points redeemable for cash. Optional alarm system to remind to take medications and attend visits.
  Arms: Novel Intervention

SUMMARY:
A randomized controlled clinical trial looking at the effect of use of a mobile phone application in addition to standard care compared to standard care alone at a youth-friendly clinic in young men who have sex with men and transgender women aged between 15-19 years at risk of HIV on PrEP adherence.

DETAILED DESCRIPTION:
OBJECTIVES

Primary Objectives:

To study PrEP adherence in adolescent MSM who are at high risk of HIV acquisition.

Secondary Objectives:

To study

1. Rates of HIV infection
2. Rates of sexually transmitted infections (STIs)
3. Sexual risk taking behaviours In adolescent MSM who are at high risk of HIV infection.

HYPOTHESES:

1. The investigators hypothesize that youth-focused interventions will produce superior adherence to PrEP from 50% with standard interventions to 70% with youth focused interventions.
2. The investigators hypothesize that adherence to PrEP varies by the level of risk behavior one perceives. Participants who take higher risk behaviors will be more likely to adhere to PrEP than participants who have lower risk behaviors. STIs are expected to be more common among participants with higher levels of adherence if they are participants who have higher risk behaviors.

RESEARCH DESIGN:

Randomised control trial, behavioural intervention

RESEARCH METHODOLOGY

1. Study population Volunteers aged 15 to under 20 years at high risk of HIV infection receiving PrEP under the 'Princess PrEP' project
2. Inclusion Criteria

   * Adolescent men who have sex with men
   * At high risk of HIV infection (have at least one of the following)

     * More than 1 sexual partner in the last 6 months
     * Irregular condom use during sexual intercourse
     * HIV positive sexual partner
   * Age 15 to under 20 years old
   * A desire to take PrEP to prevent HIV infection
   * Tested HIV negative within 1 month of enrolment
   * Able to provide written consent or assent to take part in the clinical trial
3. Exclusion criteria Signs or symptoms of acute retroviral syndrome that cannot be confirmed to be due to alternate causes, including unremitting fevers, headaches, myalgia, fatigue, and lymphadenopathy
4. Study recruitment

   * Eligible persons presenting to the Thai Red Cross Anonymous Clinic (TRCARC) or its affiliated community based organizations (Rainbow Sky Association Thailand (RSAT) Ramkamhaeng, Sex Workers in Action Group (SWING) Bangkok will be asked by counsellors on their interest to join the study.
   * Number of participants to be studied: 200
5. Informed consent process/ informed assent The research doctor will explain to potential participants about the purposes of the study and allow them to ask any questions they may have on it, and will be given time to make their decision. If a participant chooses to join the study, they will be asked for their written consent/assent and a copy of the informed consent/assent form given to them.

   * Participants aged between 15 and 18 will be asked for assent. As this is a study on sexual health where disease prevention is of utmost concern, parental consent will not be asked for.
   * Participants aged 18 to 19 will be asked for consent.
6. Study procedure After informed consent or assent, all youth will commence once daily TFV/FTC 200/300mg. Volunteers will be randomized into arms 1 (standard intervention) or 2 (novel intervention strategy). Both groups will receive youth-focused counselling by trained counsellors and have access to an adolescent-friendly sexual health promotion website and social media page where they can get in contact with counsellors, doctors, fellow adolescents and function as a platform through which they can learn about good sexual health practices. Adolescents in arm 2 (novel intervention strategy) will also receive access to a mobile phone application.

Youth-focused counselling Counsellors will provide counselling that is friendly, non-judgmental and utilize motivational interviewing techniques where sessions are more collaborative rather than didactic.

Mobile Phone Application

* Password protection will ensure user privacy
* Will allow users to input weekly data on their:

  * Sexual risk e.g. no sexual activity, sex with condoms, sex without condoms
  * PrEP use e.g. whether or not participants take their PrEP
* The application will calculate a percentage of protection users have based on their data entry
* Points can be accumulated for application use, data input to the application, for attending appointments and also for normal STI and HIV screening results. Points can be redeemed for cash
* The overall goal of the application is to increase participant awareness of self-risk and motivation to protect themselves against HIV and STI infection

Participants will be followed up at months 1, 3 and 6. At each visit, participants will complete a questionnaire on drug adherence and sexual health risk behaviours.

STI testing will be done as an indirect marker of condom use at visits 1 and 6. This will involve blood testing for syphilis serology and nucleic acid amplification testing for gonorrhea, and chlamydia on swab samples.

HIV testing will be done at all visits. TFV-DP DBS will be done at months 1, 3 and 6 to look at correlation of self-reported and actual measured PrEP compliance.

Drug Concentrations will be measured using the TFV-DP DBS at the Program for HIV Prevention and Treatment (PHPT), Chiang Mai. TFV-DP DBS levels ≥ 700 fmol/punch will be taken as adherence

ELIGIBILITY:
Inclusion Criteria:

* Adolescent men who have sex with men
* At high risk of HIV infection (have at least one of the following)

  * More than 1 sexual partner in the last 6 months
  * Irregular condom use during sexual intercourse
  * HIV positive sexual partner
* Age 15 to under 20 years old
* A desire to take PrEP to prevent HIV infection
* Tested HIV negative within 1 month of enrolment
* Able to provide written consent or assent to take part in the clinical trial

Exclusion Criteria:

* Signs or symptoms of acute retroviral syndrome that cannot be confirmed to be due to alternate causes, including unremitting fevers, headaches, myalgia, fatigue, and lymphadenopathy

Ages: 15 Years to 19 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — men who have sex with men or transgender women
Enrollment: 200 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-12-15 (Actual); Study Completion 2019-12-15 (Actual)

PRIMARY OUTCOMES:
PrEP Adherence | Weekly self-reported adherence for a period of 6 months following randomization
  Self-Reported Adherence
PrEP Adherence at 3 months | Measured at month 3 (measure of 17 day half life of TDF-DP)
  Measured Serum TDF-DP Level (from dried blood spots)
PrEP Adherence at 6 months | Measured at month 6 (measure of 17 day half life of TDF-DP)
  Measured Serum TDF-DP Level (from dried blood spots)

SECONDARY OUTCOMES:
HIV infection rates | duration of study (6 months)
  seroconversion rates whilst on PrEP during study
Rates of Urethral Neisseria gonorrhea | duration of study (6 months)
  Rates of Urethral Neisseria gonorrhea via Nucleic Acid Amplification Screening (NAAT) urine testing
Behaviour Risk-Taking | duration of study (6 months)
  Composite calculated score of risk taking based on self-reported condom use, PrEP tablets taking, number of sexual partners in preceding one month. Scores will equate to risk levels of low, medium, high and very high.
Rates of Anal Neisseria gonorrhea | duration of study (6 months)
  Rates of Anal Neisseria gonorrhea via Nucleic Acid Amplification Screening (NAAT) from anal swab samples
Rates of Urethral Chlamydia trachomatis | duration of study (6 months)
  Rates of Urethral Chlamydia trachomatis via Nucleic Acid Amplification Screening (NAAT) urine testing
Rates of Anal Chlamydia trachomatis | duration of study (6 months)
  Rates of Anal Chlamydia trachomatis via Nucleic Acid Amplification Screening (NAAT) from anal swab samples
Rates of Syphilis Infection | duration of study (6 months)
  Rates of positive treponemal blood tests
Rates of Hepatitis B infection | At initial project visit (month 0)
  Rates of positive HbsAg blood tests

CONTACTS AND LOCATIONS:
Locations (1):
- Thai Red Cross AIDS Research Center, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kawichai S, Songtaweesin WN, Wongharn P, Phanuphak N, Cressey TR, Moonwong J, Vasinonta A, Saisaengjan C, Chinbunchorn T, Puthanakit T. A Mobile Phone App to Support Adherence to Daily HIV Pre-exposure Prophylaxis Engagement Among Young Men Who Have Sex With Men and Transgender Women Aged 15 to 19 Years in Thailand: Pilot Randomized Controlled Trial. JMIR Mhealth Uhealth. 2022 Apr 21;10(4):e25561. doi: 10.2196/25561. PMID 35451976
- [Derived] Songtaweesin WN, Kawichai S, Phanuphak N, Cressey TR, Wongharn P, Saisaengjan C, Chinbunchorn T, Janyam S, Linjongrat D, Puthanakit T; CE-PID - TRC Adolescent Study Team. Youth-friendly services and a mobile phone application to promote adherence to pre-exposure prophylaxis among adolescent men who have sex with men and transgender women at-risk for HIV in Thailand: a randomized control trial. J Int AIDS Soc. 2020 Sep;23 Suppl 5(Suppl 5):e25564. doi: 10.1002/jia2.25564. PMID 32869511